CLINICAL TRIAL: NCT06299644
Title: Endoscopic Sleeve Gastroplasty Technique Comparison for Weight Loss Using the Endomina Plicating Device: A Randomized Trial
Brief Title: Endoscopic Sleeve Gastroplasty Technique Comparison for Weight Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Endo Tools Therapeutics S.A. (Industry)
Responsible Party: Principal Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P003282
Record Dates: First submitted 2024-02-01; First posted 2024-03-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Obesity, Morbid; Metabolic Disease; Weight, Body
Keywords: Endoscopic Bariatric and Metabolic Therapies (EBMT); Endoscopic Bariatric Therapies (EBT); Gastric emptying; Endoscopic Suturing; endoscopic sleeve gastroplasty (ESG); Weight Loss; Bariatric Endoscopy; Weight Management; Endoscopic plication; Gastric plication
MeSH Terms: conditions — Obesity; Obesity, Morbid; Metabolic Diseases; Body Weight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Belt and Suspenders Configuration (Active Comparator): Endoscopic sleeve gastroplasty with the Endomina system creating proximal and distal gastric plications (belt and suspenders configuration).
  Interventions: Device: Endoscopic Sleeve Gastroplasty - Belt and Suspenders
- Belt Configuration (Active Comparator): Endoscopic sleeve gastroplasty with the Endomina system creating distal gastric plications (belt configuration).
  Interventions: Device: Endoscopic Sleeve Gastroplasty - Belt

INTERVENTIONS:
Device: Endoscopic Sleeve Gastroplasty - Belt and Suspenders — Endoscopic sleeve gastroplasty using belt and suspender plications.
  Other Names: Belt and Suspenders ESG
  Arms: Belt and Suspenders Configuration
Device: Endoscopic Sleeve Gastroplasty - Belt — Endoscopic sleeve gastroplasty using belt only plications.
  Other Names: Belt ESG
  Arms: Belt Configuration

SUMMARY:
The Investigators propose suture plication placement at the distal gastric body drives a significant portion of weight loss in endoscopic sleeve and sutures only need to be placed in the distal gastric body. Therefore, in this pilot study, the investigators aim to compare "belt" with "belt and suspenders" plication pattern using the Endomina system to determine percent total weight loss.

DETAILED DESCRIPTION:
Obesity is a major global health concern. In the US, from 1999 through 2020, the prevalence of obesity has increased from 30.5% to 41.9%. Obesity, defined as the body mass index of more than 30 kg/m2, increases the risk of metabolic diseases and has become the leading cause of death including cardiovascular disease, stroke and cancers.

At present, obesity treatment ranges from lifestyle modification, pharmacotherapy, endoscopic to surgical intervention. Though bariatric surgery has proven to be the most effective treatment in terms of weight loss, it still carries the complication rates of 0.6% - 4.9%.

Endoscopic Bariatric and Metabolic Therapy (EBMT) has emerged as an alternative minimally invasive approach for the patients with morbid obesity with the body mass index (BMI) of 30 - 40 kg/m2. Endoscopic sleeve gastroplasty (ESG) involves placing sutures inside the stomach using an endoluminal full-thickness suturing device. This allows for gastric volume reduction and impaired gastric motility, which results in weight loss. Recent meta-analysis demonstrated ESG, using OverStitch suturing device, percent total weight loss (%TWL) of 16.09 - 16.43% at 12 months after procedure and a serious adverse event rate of 1 - 2.26%. With favorable outcomes and lower complication rates compared to bariatric surgery, ESG has been growing in popularity and increasingly performed worldwide. Other EBT cleared by the U.S. Food and Drug Administration for full thickness tissue approximation include the Incisionless Operating Platform endoscopic plication (USGI Medical, San Clemente, Calif, USA), and Endomina® (Endo Tools Therapeutic, Gosselies, Belgium) which creates gastric plications.

Currently, there is no standardization regarding suturing patterns. One suture pattern for gastric plication that has been used is the "belt and suspenders" pattern whereby plications sutures are placed in the distal gastric body along the width (belt) and mid/proximal gastric body (suspenders). This allows for gastric shortening and reduction in gastric volume. It is suspected this would also alter gastric motility. The distal gastric plications placed near the antrum would result in a disruption of gastric motility; decreased gastric motility would result in decrease gastric emptying and longer satiety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 18-65 years of age
2. BMI ≥ 30 kg/m2
3. Capable of giving informed consent and available to return for follow-up visit

Exclusion Criteria:

1. Untreated H. pylori infection
2. Active gastric or duodenal ulceration
3. Malignant or premalignant gastric diseases (such as intestinal metaplasia, high grade dysplasia, gastric adenocarcinoma, or gastrointestinal stromal tumor (GIST))
4. Severe reflux esophagitis (Los Angeles Classification (LA) Grade C or D)
5. Esophageal or gastric varices and/or portal hypertensive gastropathy
6. Gastroparesis
7. History of gastric surgery/endoscopic procedure
8. Active psychological issues preventing participation in a lifestyle modification program
9. Known history of endocrine disorders affecting weight (uncontrolled hypothyroidism)
10. Severe coagulopathy
11. Active smoking
12. Substance abuse
13. Serious health condition that increased risk of anesthesia and/or endoscopic procedure
14. Pregnancy or lactation
15. Patients who require Non-Steroidal Anti-inflammatory Drugs (NSAID) use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percent TWL (%TWL) | Baseline, 6 months, 12 months
  Change in the percent total weight loss from baseline at 6 and 12 months.
Adverse Events | 6 months, 12 months
  Presence of adverse events that develop post-procedure

SECONDARY OUTCOMES:
Gastric Emptying | Baseline, 6 month, 12 months
  Comparison of gastric emptying rate using Gastric Emptying Breath Test (GEBT) from baseline to 6 months and 12 months post-procedure
Number of participants with improvement in fasting glucose | Baseline, 6 months, 12 months
  Change in fasting glucose laboratory values from baseline at 6 and 12 months post-procedure
Number of participants with improvement in Hemoglobin A1c (HgA1c %) | Baseline, 6 months, 12 months
  Change in HgA1c laboratory values from baseline at 6 and 12 months post-procedure
Improvement in fasting lipids profile | Baseline, 6 months, 12 months
  Change in fasting lipids laboratory values from baseline at 6 and 12 months post-procedure
Number of participants with a change in ghrelin hormone values | Baseline, 6 months, 12 months
  Change in ghrelin laboratory values from baseline at 6 and 12 months post-procedure
Obesity-related comorbidities - hypertension | Baseline, 6 months, 12 months
  Change in hypertension diagnosis/status via change in blood pressure measurements (systolic and diastolic mm Hg) at 6 months and 12 months from baseline
Obesity-related comorbidities - change in hypertension concomitant medications | Baseline, 6 months, 12 months
  Change in hypertension diagnosis/status via change blood pressure related medication dosage (mg) at 6 months and 12 months from baseline
Obesity-related comorbidities - change in pre-diabetes/diabetes concomitant medications | Baseline, 6 months, 12 months
  Change in diabetes/pre-diabetes diagnosis/status via change in diabetes medications dosages (mg) at 6 months and 12 months from baseline
Obesity-related comorbidities - pre-diabetes/diabetes | Baseline, 6 months, 12 months
  Change in diabetes/pre-diabetes diagnosis/status via change in HgA1c measurements (%) at 6 months and 12 months from baseline
Obesity-related comorbidities - gastroesophageal reflux (GERD) | Baseline, 6 months, 12 months
  Change in GERD diagnosis/status via change in proton pump inhibitor (PPI) or related medications for treatment of GERD at 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C Thompson, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers upon written request to the PI. If PI approves of the research plan, data will be released after an Institutional Data Sharing Agreement is in place.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 months after publication of results. Available for 10 years.
Access Criteria: Formal written request to PI with research proposal/plan.

REFERENCES:
- [Background] Ibrahim AM, Ghaferi AA, Thumma JR, Dimick JB. Variation in Outcomes at Bariatric Surgery Centers of Excellence. JAMA Surg. 2017 Jul 1;152(7):629-636. doi: 10.1001/jamasurg.2017.0542. PMID 28445566
- [Background] Docimo S Jr, Aylward L, Albaugh VL, Afaneh C, El Djouzi S, Ali M, Altieri MS, Carter J; American Society for Metabolic and Bariatric Surgery Clinical Issues Committee. Endoscopic sleeve gastroplasty and its role in the treatment of obesity: a systematic review. Surg Obes Relat Dis. 2023 Nov;19(11):1205-1218. doi: 10.1016/j.soard.2023.08.020. Epub 2023 Sep 16. No abstract available. PMID 37813705
- [Background] Singh S, Hourneaux de Moura DT, Khan A, Bilal M, Ryan MB, Thompson CC. Safety and efficacy of endoscopic sleeve gastroplasty worldwide for treatment of obesity: a systematic review and meta-analysis. Surg Obes Relat Dis. 2020 Feb;16(2):340-351. doi: 10.1016/j.soard.2019.11.012. Epub 2019 Dec 10. PMID 31932205
- [Background] Li P, Ma B, Gong S, Zhang X, Li W. Efficacy and safety of endoscopic sleeve gastroplasty for obesity patients: a meta-analysis. Surg Endosc. 2020 Mar;34(3):1253-1260. doi: 10.1007/s00464-019-06889-6. Epub 2019 Jun 24. PMID 31236722
- [Background] Beran A, Matar R, Jaruvongvanich V, Rapaka BB, Alalwan A, Portela R, Ghanem O, Dayyeh BKA. Comparative Effectiveness and Safety Between Endoscopic Sleeve Gastroplasty and Laparoscopic Sleeve Gastrectomy: a Meta-analysis of 6775 Individuals with Obesity. Obes Surg. 2022 Nov;32(11):3504-3512. doi: 10.1007/s11695-022-06254-y. Epub 2022 Sep 2. PMID 36053446
- [Background] Jalal MA, Cheng Q, Edye MB. Systematic Review and Meta-Analysis of Endoscopic Sleeve Gastroplasty with Comparison to Laparoscopic Sleeve Gastrectomy. Obes Surg. 2020 Jul;30(7):2754-2762. doi: 10.1007/s11695-020-04591-4. PMID 32304011